CLINICAL TRIAL: NCT00063765
Title: A Phase I Study of NT-501-10 and NT-501-6A.02, Implants of Encapsulated Human NTC-210 Cells Releasing Ciliary Neurotrophic Factor (CNTF), in Patients With Retinitis Pigmentosa
Brief Title: Evaluation of Safety of Ciliary Neurotrophic Factor Implants in the Eye
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030234; 03-EI-0234
Record Dates: First submitted 2003-07-03; First posted 2003-07-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-03

CONDITIONS: Retinitis Pigmentosa
Keywords: NT-501; CNTF; Retinitis Pigmentosa; RP
MeSH Terms: conditions — Retinitis Pigmentosa

INTERVENTIONS:
Drug: Ciliary Neurotrophic Factor Implant NT-501

SUMMARY:
This study will evaluate the safety of a ciliary neurotrophic factor (CNTF) implant placed in the eye to allow the release of CNTF directly on the retina. The results of this study may lead to a larger investigation of CNTF implants to treat retinitis pigmentosa (RP), a progressive degenerative eye disease that begins with loss of peripheral vision and night blindness and often leads to blindness in later life.

Currently, there are no effective treatments for RP. Researchers have found, however, that certain proteins, called ciliary neurotrophic factor (CNTF), can partially protect cells in the eye if given directly inside the eye. A major challenge in treating RP is to deliver medicine directly into the eye. One way to ensure that CNTF gets into the eye is to surgically place an implant inside the eye to release the protein.

Patients 18 years of age and older with retinitis pigmentosa whose visual acuity is 20/100 or worse may be eligible for this study. Candidates will be screened with a medical history, physical examination, eye examinations, and eye photographs. The eye examination includes measurement of visual acuity and eye pressure, examination of the pupils and eye movements, and examination of the lens and back of the eye. In addition, patients will have the following tests:

* Visual field test: Patients look at a central spot on a white screen and tell the examiner whenever they see a small light appear at other places on the screen.
* Electroretinogram (ERG): Electrodes are taped to the patient's forehead. Special contact lenses are placed on the eyes, similar to normal contact lenses, after the eye has been numbed with drops. The contact lenses sense small electrical signals generated by the retina. The ERG measures the electrical activity of the retina when it is stimulated by light. For the ERG recording, the patient looks inside a large, hollow, dark sphere, and sees flashes of light, first in the dark, and then with a light turned on in the sphere.
* Optical coherence tomography: This test, done with the machine used to examine the eye, measures retinal thickness by producing cross-sectional pictures of the retina.

Participants undergo surgery at the NIH Clinical Center in a 30-minute operation to place the implant in one eye. The surgery is done under local anesthetic. Before the procedure, patients are given a steroid injection along side the eye to minimize inflammation after surgery. Following the procedure, patients return for follow-up visits once a month for 6 months. At these visits, several of the exams described above are repeated to evaluate treatment effects and check for adverse side effects. After 6 months, the implant is surgically removed. Post-surgical care for both implant and explant surgeries include examinations the day and week after surgery to examine the wound, a high dose of steroid immediately after surgery, oral antibiotics for 7 days, and eye drops for 1 week to prevent infection and inflammation.

DETAILED DESCRIPTION:
Retinitis Pigmentosa (RP) is a group of incurable degenerative diseases of the retina that have a complex molecular etiology. Approximately 100,000 Americans suffer from inherited retinal degenerative RP. More than 100 RP-inducing mutations have been identified in several genes including: rhodopsin, the rod visual pigment; peripherin, a membrane structure protein; and PDEB, the beta subunit of rod cyclic GMP (cGMP) phosphodiesterase. However, the genotype is unknown for the majority of patients. Despite this genetic heterogeneity, there tends to be a common pattern of visual loss in patients with RP. Typically, patients experience disturbance in night vision early in life due to the degeneration of rod photoreceptors. The remaining cone photoreceptors become their mainstay of vision, but over the years and decades, the cones slowly degenerate, leading to blindness. These two phases of degeneration in the visual life of an RP patient may involve different underlying pathogenic mechanisms. Regardless of the initial causative defects, the end results are photoreceptor degeneration. This common pathogenesis pathway provides a target for therapeutic intervention.

To date, there are few available, effective treatments for retinal degenerative disorders. One major challenge is to deliver potential therapeutic agents to the back of the eye, in particular to the retina. The blood-eye barrier prevents the penetration of a variety of molecules to the neurosensory retina in a similar manner to the action of the blood-brain barrier, which exists between the central nervous system and systemic circulation. To overcome this challenge, Neurotech USA, Inc. (Neurotech) developed encapsulated cell technology (ECT), specifically the NT-501-10 and NT-501-6A.02 devices, to enable controlled, sustained delivery of therapeutic agents directly into the intra-ocular fluids and thus providing direct access to the retina. ECT utilizes cells encapsulated within a semi-permeable polymer device that secretes therapeutic factors directly into the vitreous. In addition, ECT devices can be retrieved, providing an added level of safety.

Histopathologic studies have demonstrated the possibility of growth factors, neurotrophic factors, and cytokines as therapeutics for RP. Specifically, ciliary neurotrophic factor (CNTF) has proven to be the most effective in reducing retinal degeneration. Therefore, the use of implanted NT-501-10 and NT-501-6A.02 devices, which secrete CNTF into the retina, may be beneficial in patients with RP and other retinal degenerative diseases.

This pilot study will assess the ophthalmic and systemic safety, and to some extent efficacy, of the novel intra-ocular NT-501-10 and NT-501-6A.02 implants in patients with RP and poor visual acuity in one eye. The main purpose of the study is to assess the safety of the NT-501-10 and NT-501-6A.02 implants. Secondary outcomes will include the anterior chamber cell scale and vitreous haze grading to measure inflammation, which may be caused by the implant. Other secondary outcome measures related to potential product performance are visual acuity, visual fields, electroretinograms (ERG), and optical coherence tomography (OCT3) to determine retinal thickness.

ELIGIBILITY:
INCLUSION CRITERIA:

1. To participate in this study, the participant must understand and sign the protocol's informed consent (if the participant's vision is impaired to the point where it is not possible to read the informed consent document, the informed consent document will be read in its entirety to the participant).
2. Paticipant diagnosis consistent with retinitis pigmentosa (RP) characterized by the following features:

   1. progressive photoreceptor dysfunction an death
   2. clinical degeneration of the outer retina
   3. intraretinal 'bone-spicule' pigment
   4. visual field constriction
   5. night blindness
   6. major reduction of both rod and cone electroretinogram (ERG) responses.
3. The first two participants have 20/400 vision or worse in the implant (study) eye with the same or better in the fellow eye, while the remainder of the participants will have visual acuity of 20/100 or worse.
4. Participant has an ERG less than 2 MV(28-32 Hz flicker)
5. Participant with central visual field of 40 degrees diameter or less with the Goldmann V 4e stimulus (independent of a peripheral crescent of any size)
6. Participant medically able to undergo ophthalmic surgery.

EXCLUSION CRITERIA:

1. Participant less than 18 years of age.
2. Participant medically unable to comply with study procedures or follow-up visits.
3. Participant has glaucoma.
4. Participant is receiving oral or other insulin treatment for diabetes.
5. Participant has cataract and it interferes with the assessment of the posterior segment inflammation using a standard slit lamp examination.
6. Participant has undergone intra-ocular lens replacement less than 6 months prior to enrollment.
7. Participant has participated in any other clinical trial of a drug or device within the last 6 months.
8. Participant is on chemotherapy.
9. Participant is on ocular medications known to be toxic to the lens, retina, or optic nerve.
10. Participant who is pregnant.
11. Participant with retinal inflammatory diseases.
12. Participant with macula edema
13. Participant with history of malignancy (except study participants having a basal cell carcinoma that was treated successfully, or other malignancy operated on and in remission of 5 years prior to inclusion in the trial).
14. Participant is considered immunodeficient or has a known history of HIV.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2003-06; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Aebischer P, Schluep M, Deglon N, Joseph JM, Hirt L, Heyd B, Goddard M, Hammang JP, Zurn AD, Kato AC, Regli F, Baetge EE. Intrathecal delivery of CNTF using encapsulated genetically modified xenogeneic cells in amyotrophic lateral sclerosis patients. Nat Med. 1996 Jun;2(6):696-9. doi: 10.1038/nm0696-696. PMID 8640564
- [Background] Aebischer P, Kato AC. Treatment of amyotrophic lateral sclerosis using a gene therapy approach. Eur Neurol. 1995;35(2):65-8. doi: 10.1159/000117095. PMID 7796839
- [Background] A phase I study of recombinant human ciliary neurotrophic factor (rHCNTF) in patients with amyotrophic lateral sclerosis. The ALS CNTF Treatment Study (ACTS) Phase I-II Study Group. Clin Neuropharmacol. 1995 Dec;18(6):515-32. doi: 10.1097/00002826-199512000-00004. PMID 8681312
- [Derived] Kauper K, McGovern C, Sherman S, Heatherton P, Rapoza R, Stabila P, Dean B, Lee A, Borges S, Bouchard B, Tao W. Two-year intraocular delivery of ciliary neurotrophic factor by encapsulated cell technology implants in patients with chronic retinal degenerative diseases. Invest Ophthalmol Vis Sci. 2012 Nov 1;53(12):7484-91. doi: 10.1167/iovs.12-9970. PMID 23049090